CLINICAL TRIAL: NCT05735847
Title: Does Surgery-Induced Trauma Influence Postoperative Safety and Outcome Comparing Total vs. Medial Unicompartmental Knee Arthroplasty (SITA): A Prospective Cohort Study
Brief Title: Surgery Induced Trauma After Total Versus Medial Unicompartmental Knee Arthroplasty (SITA)
Acronym: SITA
Status: Active, not recruiting | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Frederiksberg University Hospital (Other); Parker Research Institute (Other)
Responsible Party: Principal Investigator, Anders Troelsen, Head of Clinical Orthopaedic Surgery Hvidovre (CORH), Clinical Professor, Hvidovre University Hospital
Other Study IDs: H-22029746
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis; Arthritis; Surgery; Total Knee Arthroplasty; Unicompartmental Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CRP, Interleukin-1-beta(IL1-beta), interleukin-6 (IL6), Interleukin-8(IL8), tumor necrosis factor alfa (TNF-alfa), Metalloproteinases (MMP3, MMP9, MMP13), calprotectin - S100 calcium binding protein A8/A9 (S100A8/S100A9), S100 calcium-binding protein B (S100B), CRP, Haemoglobin (Hb), Erytrocyte Sedimentation Rate (ESR), White cell count (L+D), Platelets, Myoglobin, Lactate dehydrogenase (LDH), Creatine Kinase (CK).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total Knee Arhroplasty (TKA): Study participants will be adults (i.e. at least 18 years old) who have diagnosis of KOA with an indication for primary Total Knee Arthroplasty (TKA).
  Interventions: Procedure: Total Knee Arthroplasty (TKA)
- Unicompartmental Knee Arthroplasty (UKA): Study participants will be adults (i.e. at least 18 years old) who have diagnosis of KOA with an indication for primary medial Unicompartmental Knee Arthroplasty (UKA).
  Interventions: Procedure: Unicompartmental Knee Arthroplasty (UKA)

INTERVENTIONS:
Procedure: Total Knee Arthroplasty (TKA) — The choice between TKA and UKA is based on the radiological presentation of the knee KOA on an x-ray. A surgery with TKA involves the replacement of both the medial and lateral compartments of the knee.
  Groups: Total Knee Arhroplasty (TKA)
Procedure: Unicompartmental Knee Arthroplasty (UKA) — The choice between TKA and UKA is based on the radiological presentation of the knee KOA on an x-ray. A surgery with UKA involves the replacement of one compartment.
  Groups: Unicompartmental Knee Arthroplasty (UKA)

SUMMARY:
Osteoarthritis (OA) is the most common type of arthritis, characterized by pain and physical disability. More than 10% of persons > 55 years have symptomatic OA, primarily involving the knees. Knee arthroplasty is considered a successful orthopaedic procedure in progressed knee OA (KOA) with severe pain and disability where non-surgical treatments have been tried.

It has long been recognized that injury to the body, either from trauma or surgery causes an inflammatory response. As TKA is considered a more invasive procedure compared with UKA, TKA and UKA may not trigger inflammatory reactions of the same magnitude. Differences in inflammatory response between TKA and UKA could help explain why differences in outcome are present, despite both procedures being technically successful.

Even though knee arthroplasty is a very common and successful procedure, there are no existing studies comparing the invasiveness of TKA and UKA. As morbidity and mortality rates differ between the groups, the aim of this prospective cohort study is to investigate whether the post-operative inflammatory responses differ between TKA and UKA, and secondarily whether this difference can explain the difference in outcome between the two procedures.

The investigators hypothesize that TKA generates a larger postoperative systemic inflammatory response compared with UKA due to more extensive periarticular soft tissue and bone trauma.

The study's primary outcome is C-reactive Protein (CRP) measured in blood 24 hours after surgery (22-26 hours after surgery ~ day 1).

Participants which are candidates for either a TKA or a UKA will through serial blood test measurement have their postoperative systemic inflammatory response measured. This further will be correlated to the clinical and functional outcomes over a 2-years postoperative follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more
* A clinical and radiological diagnosis of knee OA
* Candidate for spinal anaesthesia
* signed informed consent

Exclusion Criteria:

* Planned surgery within the observation period other than KA
* Any contraindications to the use of torniquet during surgery
* Any contraindication to the administration of pre-operative dexamethasone
* KA indication due to sequelae of e.g. fracture(s)
* Previous infection of the target knee joint
* Injection of medication or substances in the target knee within 3 months prior to participation
* Immuno-inflammatory arthritis as cause of knee OA
* Known autoimmune and/or inflammatory disease e.g. colitis ulcerosa
* Active cancer diagnosis with ongoing treatment
* Current systemic treatment with glucocorticoids equivalent to > 7.5 mg prednisolone/day
* Surgery requiring spinal/general anaesthesia within the last 3 months prior to inclusion
* Infection requiring medical/surgical treatment within the last 4 weeks prior to surgery for KA
* Neurological dysfunction compromising mobility
* Inability to understand or read Danish incl. instructions and questionnaires
* Any other condition or impairment that, in the opinion of the investigator (or his/her delegate), makes a potential participant unsuitable for participation or which obstruct participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be adults (i.e. at least 18 years old) who have diagnosis of KOA with an indication for primary KA (medial unicondylar or total arthroplasty).
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
C-reactive protein (CRP) | Day 1 (24 hours after surgery)
  Marker of systemic inflammation and soft tissue injury

SECONDARY OUTCOMES:
Interleukin-1-beta (IL1-beta) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
Interleukin-6 (IL6) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
Interleukin-8 (IL8) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
Tumor necrosis factor alfa (TNF-alfa) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
Metalloproteinases (MMP3, MMP9, MMP13) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
Calprotectin - S100 calcium binding protein A8/A9 (S100A8/S100A9) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
S100 calcium-binding protein B (S100B) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
C-Reactive Protein (CRP) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
Haemoglobin (Hb) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
Erythrocyte Sedimentation Rate (ESR) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
White cell count (L+D) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
Platelets | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
Myoglobin | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
Lactate dehydrogenase (LDH) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
Creatine Kinase (CK) | Baseline, 2 hours, 1 day, 7 days, and 21 days (after surgery)
  Marker of systemic inflammation and soft tissue injury
Duration of surgery in minutes | Within the first week after surgery
  The time from when the surgeon of record starts the procedure until he/she leaves the procedure.
  This information will be collected from the patient's medical record.
Postoperative x-rays | On day of surgery, or postoperative day 1, or postoperative day 2
  Postoperative x-rays of the knee are performed routinely in order to evaluate whether implants are placed in accordance with recommendations.
Knee pain (VAS) | Day 1, day 7, day 21, 3 months, 6 months, 12 months, 24 months (after surgery)
  Pain assessed using the visual analogue score (VAS) following surgery. The Scores go from 0-10. 0 = no pain. 10 = the most pain. The patients indicate how their pain during the last 24 hours fit in to the scale.
Analgesia requirements after surgery | Day 1, day 7, day 21, 3 months (after surgery)
  Both preoperative and postoperative requirement of analgesia will be noted. Analgesia requirement will include Paracetamol, NSAID, Acetylic Acids and Opioids. Type of anaesthesia/sedation used during surgery will in addition be recorded. The above information will be collected from the patient's medical record.
Perioperative complications | 1 day During admission (after surgery)
  Complications which happens during surgery.
Length of stay/ Re-admissions within the first 90 days | 90 days (after surgery)
  The patients are expected to be discharged on day 1 post-surgery after a blood sample is taken at 24 hours post-surgery. It will be recorded if a patient is not able to be discharged at this time and for how many days the admission will last. The number of readmissions within 90 days of surgery and the reason for re-admission will also be recorded. This information will be collected from the patient's medical journal.
90 days complications (medical, surgical) | 90 days (after surgery)
  Complications (both medical and surgical) arising within 90 days of surgery will be recorded. The information will be collected from the patient's medical records.
  Complications includes myocardial infarction/cardiac events, cerebrovascular events, venous thromboembolism, deep infection, reoperation, revision, and death.
Data on any revisions performed on includes patient within 24 months | 24 months (after surgery)
  Any revisions in patients within 24 months will be recorded. The reason for revision and the type of revision will be noted. The information will be collected from the patient's medical records.
Pain Catastrophizing Scale (PCS) | Baseline
  The Pain Catastrophizing Scale (PCS) is a 13-item patient reported outcome measure developed to evaluate catastrophic thinking related to pain. Standardized answer options are given through a 5-point Likert scales, from 0 (not at all) to 4 (all the time). Higher scores indicate higher level of catastrophizing. A total score yielding (ranging from 0-52), along with three subscale scores assessing rumination, magnification, and helplessness.
Pain Detect Questionnaire (PDQ) | Baseline
  The PDQ is a patient administered questionnaire used to assess the likelihood of a pain experience being of neuropathic origin.
Oxford Knee Score (OKS) | Baseline, 3 months, 6 months, 12 months, 24 months (after surgery)
  The Oxford Knee Score (OKS) is a 12-item patient reported outcome questionnaire developed specifically to assess the patient's perspective on the outcomes of knee arthroplasty with respect to combined pain and physical function. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. Thus, a total score is calculated from 0 to 48, with 48 indication the best outcome. The OKS is short, practical, reliable, valid, and sensitive to clinically important changes over time18.
The Forgotten Joint Score | Baseline, 3 months, 6 months, 12 months, 24 months (after surgery)
  The Forgotten Joint Score was designed to assess patient outcome in patients undergoing conservative or operative treatment of the knee, and it analyses patient's ability to forget about a joint as a result of successful treatment. The questionnaire consists of 12 questions that are equally weighted and measure patient satisfaction. Standardized answer options are given (6 Likert boxes). Scores are summed to create a composite score that is converted to a 100-point scale. Higher scores indicate greater satisfaction.
European Quality of Life questionnaire with 5 dimensions for adults (EQ-5D) | Baseline, 3 months, 6 months, 12 months, 24 months (after surgery)
  EQ-5D-5L is a standardized patient-reported instrument for measurement of health outcome and quality of life. EQ-5D-5L is designed for self-completion by respondents and is ideally suited for use in surveys. The EQ-5D-5L consists of 2 pages - the EQ-5D-5L description system and the EQ Visual Analogue Scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Standardized answer options are given (5 22.12.2022 Page 17 of 30 Likert boxes) and each question is assigned a score from 1 to 5. Instructions to respondents are included in the questionnaire. The EQ VAS records the respondent's self-rated health on a 20 visual analogue scale with endpoints labelled "the best health you can imagine" and "the worst health you can imagine". This information can be used as a quantitative measure of health judged by the individual respondents.
Patient acceptable Symptom States (PASS) | 3 months, 6 months, 12 months, 24 months (after surgery)
  One question regarding PASS will be used to assess how many patients consider themselves well after surgery (as opposed to feeling better). PASS is assessed as a dichotomous outcome (yes/no) to the question:"Taking into account all the activities you have during your daily life, your level of pain, and also your functional impairment, do you consider that your current state is satisfactory?". The actual question asked will be in Danish (Appendix G).
Treatment failure (TF) | 3 months, 6 months, 12 months, 24 months (after surgery)
  We will define treatment failure in two ways:
  1. Patients replying 'no' to the PASS question (above) will be asked to answer (yes/no) the following question: "Would you consider your current state as being so unsatisfactory that you think the treatment has failed?" Patients replying, 'yes' to this second question will be defined as experiencing 'treatment failure' (TF).
  2. Patients who during the observation period undergo revision surgery are defined as TF. We will seek information about the reason for revision surgery (e.g. infection, malalignment, loosening/lysis, implant wear, dislocation/instability, stiffness, pain, and other reasons) in the medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Troelsen, MD, PhD, DMSc, Principal Investigator — Department of Orthopaedic Surgery, Amager Hvidovre Hospital, Kettegård Alle 30, DK-2650 Hvidovre
Locations (1):
- Department of Orthopaedic Surgery, Amager Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan